CLINICAL TRIAL: NCT04118088
Title: Postauthorization Safety Study of the Long-Term Safety and Efficacy of Repeat Administration of Darvadstrocel in Patients With Crohn's Disease and Complex Perianal Fistula
Brief Title: A Study of Darvadstrocel in Adults With Crohn's Disease and Complex Perianal Fistula
Acronym: EMPIRE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alofisel-4001; EUPAS31439 (Registry Identifier: ENCePP); 2022-503014-23-00 (EU CTIS Number); 2017-002491-10 (EudraCT Number)
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease; Complex Perianal Fistula
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Darvadstrocel (Experimental): Participants who had previously received darvadstrocel were administered a single repeat dose of darvadstrocel, 24 mililiter (mL) suspension of 120 million cells (5 million cells/mL), as a perilesional injection into the fistula.
  Interventions: Biological: Darvadstrocel

INTERVENTIONS:
Biological: Darvadstrocel — Darvadstrocel suspension of human expanded adipose stem cells.
  Other Names: Alofisel; Cx601

SUMMARY:
The main aim is to check the long term side effects of a repeat treatment of darvadstrocel and to see if that treatment improves symptoms of Crohn's disease and complex perianal fistula. Participants will attend 8 clinic visits and will receive 1 treatment of darvadstrocel at the third visit. A magnetic resonance imaging (MRI) will be performed several times during the study.

DETAILED DESCRIPTION:
The biological being tested in this study is called darvadstrocel (Alofisel). This study is examining the long-term safety and efficacy of a repeat dose of darvadstrocel in people who have Crohn's disease and complex perianal fistula.

The study will enroll approximately 50 patients. Participants will be assigned to one treatment group to receive:

• Darvadstrocel 120 million cells

All participants would be allowed to receive one repeat dose of darvadstrocel in the whole study. This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 3 years. Participants will make multiple visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, ICF and any required privacy authorization before the initiation of any study procedures.
3. The participant is male or female and aged 18 years or older.
4. The participant has complex perianal fistula(s) with a maximum of 2 internal openings and a maximum of 3 external openings based on clinical assessment and a reading of a locally-performed contrast enhanced (gadolinium) pelvic MRI. Fistula(s) must have been draining for at least 6 weeks prior to baseline visit. A complex perianal fistula is defined as a fistula that meets 1 or more of the following criteria:

   1. High inter-sphincteric, high trans-sphincteric, extra-sphincteric or suprasphincteric.
   2. Presence of ≥2 external openings.
   3. Associated perianal abscess(es). Note: Abscesses that are larger than 2 cm in at least 2 dimensions on MRI must be confirmed to have been drained adequately by the surgeon during the preparation curettage in order to be eligible.
5. The participant has already received treatment with darvadstrocel for a complex perianal fistula at least 6 months prior to baseline visit for retreatment, and their physician has planned a repeat treatment administration for the original tract (full remission not obtained or relapse of fistula draining) or for a new complex perianal fistula tract.
6. The participant has controlled or mildly active Crohn's disease (CD) (defined as patient reported outcomes measure derived from CDAI patient reported outcome score-2 [PRO-2] score <14).
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use barrier method of contraception (e.g. condom with or without spermicide) from signing of informed consent and until 1 year after repeat administration.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use a highly effective/effective method of contraception from signing of informed consent and until 1 year after repeat administration.

Exclusion Criteria:

1. The participant has lack of clinical response to prior treatment with darvadstrocel, where clinical response is defined as closure of at least 50% of all treated external fistula openings that were draining at baseline despite gentle finger compression or in the case of a unique fistula, a partial closure of the fistula.
2. The participant has a history of hypersensitivity or allergies to darvadstrocel or related compounds.
3. The participant has a history of hypersensitivity or allergies to penicillin or to aminoglycosides; Dulbecco modified eagle medium; bovine serum; local anesthetics or gadolinium.
4. The participant is currently participating in a double-blind clinical study with darvadstrocel. Participants participating in the ongoing INSPIRE registry (Alofisel-5003) study would need to withdraw from that study in order to enroll in this study.
5. The participant is currently receiving or has received any other investigational medicinal product (IMP) within the last 3 months or at least 5 times the respective elimination half-life time, whichever is longer, before signing the ICF.
6. The participant has known or suspected COVID-19 by the investigator within the past 2 months (additional testing may be performed at the discretion of the investigator). Positive antibody testing for COVID without other evidence of current or recent active infection does not exclude participation.

   a) Participants who were in screening at the time that COVID 19-related factors resulted in discontinuation may also be rescreened with approval of the sponsor or designee.
7. The participant has major alterations in any of the following laboratory tests:

   1. Serum creatinine levels >1.5 times the upper limit of normal (ULN).
   2. Total bilirubin >1.5 × ULN.
   3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3.0 × ULN.
   4. Hemoglobin <10.0 grams per deciliter (g/dL).
   5. Platelets <75.0 × 10^9 per liter (/L).
   6. Albumin <3.0 g/dL.
8. The participant has an increased risk for a surgical procedure.
9. The participant has a known chronically active hepatopathy of any origin, including cirrhosis and participants with persistent positive hepatitis B surface antigen and quantitative hepatitis B virus polymerase chain reaction (PCR) or positive serology for hepatitis C virus (HCV) and quantitative HCV PCR within 6 months before the baseline visit.
10. If female, the participant is pregnant or breastfeeding, or intending to become pregnant before participating in this study, during the study, or intending to donate ova during such time period.
11. If male, the participant intends to donate sperm during this study.
12. The participant has a contraindication to MRI scan (e.g., due to the presence of pacemaker, hip replacement, severe claustrophobia, or renal insufficiency as defined by local clinical guidelines).
13. The participant has a contraindication to the anesthetic procedure.
14. The participant has severe rectal and/or anal stenosis that would make it impossible to follow the surgery procedure.
15. The participant has severe proctitis (rectal ulcers >0.5 cm) that would make it impossible to follow the surgery procedure.
16. The participant has any prior invasive malignancy diagnosed within the last 3 years before baseline visit. Participants with basal cell carcinoma of the skin completely resected outside the perineal region can be included.
17. The participant has a current or recent (within 6 months before the baseline visit) history of severe, progressive, and/or uncontrolled hepatic, hematologic, gastrointestinal (other than CD), renal, endocrine, pulmonary, cardiac, neurologic, or psychiatric disease that may result in participant's increased risk from study participation and/or lack of compliance with study procedures.
18. The participant has had major surgery of the gastrointestinal tract within 6 months before baseline or any minor surgery of the gastrointestinal tract 3 months before baseline.
19. The participant had local major perianal surgery, and/or treatment with darvadstrocel within 6 months before baseline. The abscess drainage, cleaning surgery, or seton placement are not considered as "local major surgery" in this protocol.
20. The participant does not wish to or cannot comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (30):
- Akh Wien, Vienna, Austria
- Czechia (2):
  - NH Hospital a.s., Hořovice
  - ISCARE a.s., Prague
- France (7):
  - CHU de Nice - Hopital de l'Archet II - Gastro-Enterologie, Hepatologi, Nice, Alpes-Maritimes
  - CHRU Hopital de Pontchaillou - Maladies De L'Appareil Digesti, Rennes, Ille-et-Vilaine
  - CHRU de Lille - Hopital Claude Huriez - Gastroenterologie, Lille, Nord
  - CHU AMIENS PICARDIE Site SUD Hepato-Gastroenterology, Amiens, Picardie
  - Centre Hospitalier Lyon Sud - Gastroenterology, Pierre-Bénite, Rhone
  - Paris St. Joseph Hospital, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
- Germany (4):
  - Klinikum Dresden, University Hospital Dresden, Dresden, Saxony
  - Stadtisches Klinikum Luneburg, Luneburg, Schleswig-Holstein
  - Charite - Campus Benjamin Franklin, Berlin
  - Krankenhaus Waldfriede, Berlin
- Israel (5):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-Karem, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim sheba Medical Center, Tel Litwinsky
- Spain (11):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Nuestra Senora de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - H. Donostia, Donostia / San Sebastian, San Sebastian
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - C.H.U. de Pontevedra, Pontevedra
  - H.C.U. de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a35a??page=1&idFilter=Alofisel-4001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 22 December 2020 to 14 February 2025.
Pre-assignment Details: Participants with a diagnosis of Crohn's Disease (CD) and complex perianal fistula were enrolled in this study to receive a single repeated administration of darvadstrocel (Alofisel). The study was terminated early based on the sponsor's decision.
Groups:
- Darvadstrocel: Participants who had previously received darvadstrocel were administered a single repeat dose of darvadstrocel, 24 mililiters (mL) suspension of 120 million cells (5 million cells/mL), as a perilesional injection into the fistula.
Period: Overall Study
Arm/Group | Darvadstrocel
Started | 53
Completed | 11
Not Completed | 42
Not completed — Study Terminated by Sponsor | 38
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) consisted of all participants who were enrolled in the study and received treatment with darvadstrocel.
Groups:
- Darvadstrocel: Participants who had previously received darvadstrocel were administered a single repeat dose of darvadstrocel, 24 mL suspension of 120 million cells (5 million cells/mL), as a perilesional injection into the fistula.
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: From signing of informed consent form (ICF) up to 156 weeks post-repeat administration (the only administration in this study), up to approximately 164 weeks
Population: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
percentage of participants | 66

2. Primary Outcome: Percentage of Participants With at Least One Treatment Emergent Serious Adverse Event (TESAE)
Description: A serious adverse event (SAE) is defined as an untoward medical occurrence, significant hazard, contraindication, side effect or precaution that at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent SAE is an SAE which occurs after exposure to study treatment. Percentages were rounded off to the nearest single decimal place.
Time Frame: From signing of ICF up to 156 weeks post-repeat administration (the only administration in this study), up to approximately 164 weeks
Population: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
percentage of participants | 5.7

3. Primary Outcome: Number of Reported Pregnancies During Study
Description: Female participants and/or female partners of male participants who become pregnant following treatment with the study product and reported the pregnancy on a paper pregnancy report form immediately or within 24 hours of awareness were reported.
Time Frame: From administration of repeat dose up to 156 weeks post-repeat administration
Population: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel.
Measure: Number; unit: pregnancies
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
pregnancies | 1

4. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Event of Special Interest (TEAESI)
Description: Adverse event of special interests (AESIs) include immunogenicity/alloimmune reactions, hypersensitivity reactions, ectopic tissue formation, medication errors, tumorigenicity, and transmission of infectious agents. A treatment-emergent AESI is an AESI which occurs after exposure to study treatment.
Time Frame: as for outcome 2
Population: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
percentage of participants | 17

5. Secondary Outcome: Percentage of Participants Who Achieved Combined Remission of Perianal Fistula(s)
Description: Combined remission was defined as the closure of all treated external openings that were draining at baseline, despite gentle finger compression and absence of collection(s) >2 centimeters (cm) (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by central magnetic resonance imaging (MRI) assessment.
Time Frame: At Weeks 24 and 156 post-repeat darvadstrocel administration
Population: As the sponsor decided to terminate the study before the MRI could be done, the data for this outcome measure which was planned to be collected through MRI was not collected.
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission
Description: Clinical remission was defined as closure of all treated external fistula openings that were draining at baseline despite gentle finger compression.
Time Frame: At Weeks 6, 24, 52, 104, and 156 post-repeat darvadstrocel administration
Population: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel. Number analyzed is the number of participants available for analysis at the specified time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
percentage of participants
  Week 6 | 52.8 [38.6 to 66.7]
  Week 24 | 66.0 [51.7 to 78.5]
  Week 52: number analyzed (Participants) | 52
  Week 52 | 69.2 [54.9 to 81.3]
  Week 104: number analyzed (Participants) | 27
  Week 104 | 74.1 [53.7 to 88.9]
  Week 156: number analyzed (Participants) | 11
  Week 156 | 72.7 [39.0 to 94.0]

7. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response
Description: Clinical response was defined as closure of at least 50% of all treated external fistula openings that were draining at baseline despite gentle finger compression.
Time Frame: At Weeks 6, 24, 52, 104, and 156 post-repeat darvadstrocel administration
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
percentage of participants
  Week 6: number analyzed (Participants) | 52
  Week 6 | 61.5 [47.0 to 74.7]
  Week 24: number analyzed (Participants) | 52
  Week 24 | 71.2 [56.9 to 82.9]
  Week 52: number analyzed (Participants) | 52
  Week 52 | 73.1 [59.0 to 84.4]
  Week 104: number analyzed (Participants) | 27
  Week 104 | 77.8 [57.7 to 91.4]
  Week 156: number analyzed (Participants) | 11
  Week 156 | 72.7 [39.0 to 94.0]

8. Secondary Outcome: Percentage of Participants With Relapse From Week 24 Combined Remission
Description: Relapse was defined as reopening of any of the treated fistula(s) external openings with active drainage as clinically assessed that were in the combined remission at Week 24 or the development of a collection >2 cm (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by centrally read MRI assessment.
Time Frame: From Week 24 to Week 156 post-repeat darvadstrocel administration
Population: as for outcome 5
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 0

9. Secondary Outcome: Time to Relapse
Description: Time to Relapse was defined as the time in days to reopening of any of the treated fistula(s) external openings with active drainage as clinically assessed, relative to Week 24.
Time Frame: From Week 24 to the day of relapse post-repeat darvadstrocel administration
Population: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel. Time to relapse is presented in the subset of participants who were in clinical remission at Week 24.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 35
days | 932.0 [748.0 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to censoring.

10. Secondary Outcome: Percentage of Participants With New Perianal Abscess in Treated Fistula
Time Frame: At Weeks 6, 24, 52, 104, and 156 post-repeat darvadstrocel administration
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
percentage of participants
  Week 6 | 3.8
  Week 24 | 5.7
  Week 52 | 0
  Week 104 | 0
  Week 156: number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Score of Discharge and Pain Items of Perianal Disease Activity Index (PDAI) Score
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) discharge; (b) pain; (c) restriction of sexual activity; (d) type of perianal disease; and (e) degree of induration. Each item is graded on a 5-point scale ranging from no symptoms (score of 0) to severe symptoms (score of 4). Higher score means more severe disease.
Time Frame: Baseline to Weeks 6, 24, 52, 104, and 156 post-repeat darvadstrocel administration
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 53
score on a scale
  Discharge: Baseline | 1.4 (0.95)
  Discharge: Change at Week 6 | -0.3 (1.17)
  Discharge: Change at Week 24 | -0.6 (1.16)
  Discharge: Change at Week 52: number analyzed (Participants) | 52
  Discharge: Change at Week 52 | -0.6 (1.32)
  Discharge: Change at Week 104: number analyzed (Participants) | 27
  Discharge: Change at Week 104 | -0.6 (1.39)
  Discharge: Change at Week 156: number analyzed (Participants) | 11
  Discharge: Change at Week 156 | -0.4 (1.36)
  Pain Restriction of Activities: Baseline | 1.1 (0.79)
  Pain Restriction of Activities: Change at Week 6 | -0.5 (0.95)
  Pain Restriction of Activities: Change at Week 24 | -0.5 (0.93)
  Pain Restriction of Activities: Change at Week 52: number analyzed (Participants) | 52
  Pain Restriction of Activities: Change at Week 52 | -0.6 (1.00)
  Pain Restriction of Activities: Change at Week104: number analyzed (Participants) | 27
  Pain Restriction of Activities: Change at Week104 | -0.6 (0.80)
  Pain Restriction of Activities: Change at Week156: number analyzed (Participants) | 11
  Pain Restriction of Activities: Change at Week156 | -0.8 (0.87)
  Restriction of Sexual Activity: Baseline | 1.1 (1.43)
  Restriction of Sexual Activity: Change at Week 6 | -0.4 (0.99)
  Restriction of Sexual Activity: Change at Week 24 | -0.4 (1.10)
  Restriction of Sexual Activity: Change at Week 52: number analyzed (Participants) | 52
  Restriction of Sexual Activity: Change at Week 52 | -0.5 (1.23)
  Restriction of Sexual Activity: Change at Week104: number analyzed (Participants) | 27
  Restriction of Sexual Activity: Change at Week104 | -0.4 (1.31)
  Restriction of Sexual Activity: Change at Week156: number analyzed (Participants) | 11
  Restriction of Sexual Activity: Change at Week156 | -0.8 (1.25)
  Type of Perianal Disease: Baseline | 2.0 (0.48)
  Type of Perianal Disease: Change at Week 6 | -0.4 (0.88)
  Type of Perianal Disease: Change at Week 24 | -0.8 (1.11)
  Type of Perianal Disease: Change at Week 52: number analyzed (Participants) | 52
  Type of Perianal Disease: Change at Week 52 | -0.8 (1.16)
  Type of Perianal Disease: Change at Week 104: number analyzed (Participants) | 27
  Type of Perianal Disease: Change at Week 104 | -0.8 (1.24)
  Type of Perianal Disease: Change at Week 156: number analyzed (Participants) | 11
  Type of Perianal Disease: Change at Week 156 | -0.6 (0.92)
  Degree of Induration: Baseline | 1.1 (0.81)
  Degree of Induration: Change at Week 6 | -0.4 (1.03)
  Degree of Induration: Change at Week 24 | -0.5 (1.03)
  Degree of Induration: Change at Week 52: number analyzed (Participants) | 52
  Degree of Induration: Change at Week 52 | -0.7 (0.90)
  Degree of Induration: Change at Week 104: number analyzed (Participants) | 27
  Degree of Induration: Change at Week 104 | -0.6 (0.85)
  Degree of Induration: Change at Week 156: number analyzed (Participants) | 11
  Degree of Induration: Change at Week 156 | -0.5 (0.82)

ADVERSE EVENTS:
Time Frame: From signing of ICF up to 156 weeks post-repeat administration (the only administration in this study), up to approximately 164 weeks
Description: SAF consisted of all participants who were enrolled in the study and received treatment with darvadstrocel.
Arm/Group | Darvadstrocel
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 3/53
Other Adverse Events (participants affected / at risk) | 20/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darvadstrocel (N=53)
Anal abscess (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darvadstrocel (N=53)
COVID-19 (Infections and infestations) | 7
Diarrhoea (Gastrointestinal disorders) | 3
Fistula discharge (Musculoskeletal and connective tissue disorders) | 3
Influenza (Infections and infestations) | 3
Proctalgia (Gastrointestinal disorders) | 8

LIMITATIONS AND CAVEATS:
The study was terminated early based on sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT04118088/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT04118088/SAP_001.pdf